CLINICAL TRIAL: NCT06514495
Title: Differential Effects of in Vivo and Virtual Exposure Therapy on the Interoception and Reactivity of Different Body Systems in Agoraphobia
Brief Title: Differential Effects of in Vivo and Virtual Exposure Therapy in Agoraphobia
Acronym: VRExpo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Vanessa Renner, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-17625
Record Dates: First submitted 2024-07-02; First posted 2024-07-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Agoraphobia; Panic; Social Anxiety Disorder
Keywords: exposure; virtual reality; interoception; cortisol; immune system; endocannabinoids
MeSH Terms: conditions — Agoraphobia; Phobia, Social | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality exposure (Active Comparator): Agoraphobic patients receive exposure therapy in virtual reality
  Interventions: Other: Therapy
- In vivo exposure (Active Comparator): Agoraphobic patients receive exposure therapy in vivo
  Interventions: Other: Therapy

INTERVENTIONS:
Other: Therapy — Cognitive behavioral psychotherapy with exposure

SUMMARY:
Anxiety disorders, including agoraphobia, are prevalent in the German population, leading affected individuals to avoid specific places like crowds or public transport. Although cognitive-behavioral therapy with exposure is an effective treatment, many patients resort to medication rather than therapy. Virtual Reality Exposure Therapy (VRET) shows promise in easing exposure treatment with customizable scenarios. Interoception (body symptom perception) and the endocannabinoid system are explored as factors in maintaining agoraphobia. Studies investigate how therapies like exposure (both in vivo and in VR) impact these factors and treatment outcomes. Interoception, especially in panic disorder patients, plays a crucial role, with accurate heartbeat perception linked to maintaining anxiety. The endocannabinoid system, affecting various functions, is studied for its role in therapy outcomes and its modulation of the body's stress response. The study aims to understand how these systems interact in agoraphobic patients and how therapy affects their functionality.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common mental illnesses in the German population. Agoraphobia is an anxiety disorder characterized by the avoidance of specific places. Individuals affected by agoraphobia, for example, avoid crowds, public transportation, or traveling far from home, which significantly impacts their daily life. Due to the high psychological distress experienced by those affected, they often seek treatment, making agoraphobia one of the most common diagnoses in outpatient psychotherapy. Cognitive-behavioral therapy with exposure in vivo is considered the "gold standard" of psychotherapeutic treatment for agoraphobia, as it consistently shows high therapeutic effects. However, studies show that 90% of agoraphobic patients take psychotropic medication, and only 17% are in psychotherapeutic treatment. Despite the effectiveness of exposure therapy, it is rarely used in outpatient practice. Based on a survey, only 13-17% of psychotherapists conduct exposure therapy. Other studies indicate that only 8% of agoraphobic patients receive exposure therapy. Due to persistent avoidance behaviors and the limited availability of effective exposure therapy, the suffering and likelihood of chronicity of the condition increase.

Exposure therapy in virtual reality (VR) seems to offer a promising solution to this problem due to its ease of implementation compared to in vivo exposure. By programming anxiety-inducing scenarios for agoraphobic patients in VR, exposure could be conducted with less time and cost. Additionally, it offers other benefits such as the individual customization of anxiety-inducing scenarios. Various studies have already demonstrated the effectiveness of Virtual Reality Exposure Therapy (VRET) in treating various anxiety disorders. In agoraphobic patients, significant reductions in subjectively reported symptoms have been observed, as well as an impact of VRET on psychophysiological measures (e.g., electrodermal activity) indicating physiological arousal during exposure. Both in vivo exposure and VR exposure lead to a reduction in subjective symptoms in agoraphobic patients, and initial effects on psychophysiological parameters (e.g., heart rate variability) have been demonstrated.

Despite the positive effects of in vivo exposure therapy and VRET, agoraphobic symptoms often persist after psychotherapeutic treatment or there is a recurrence of symptoms after initial improvement. Previous studies have identified various factors that could contribute to maintaining the symptoms. In the planned study, interoception and the function of different body systems are the focus as maintaining factors of agoraphobia. It will be investigated how these factors influence treatment outcomes and are influenced by exposure therapies (in vivo vs. VR).

Interception as a maintaining factor of agoraphobia Interoception, the perception of body symptoms, plays a key role in cognitive-behavioral models of mental disorders. In patients with panic disorder (PD), it has been found that they have more accurate cardiac interoceptive rates than healthy controls. Specifically, it has been shown that good heartbeat perception is associated with high relapse rates. In the context of panic attacks, more accurate perception of a rapid heartbeat could contribute to maintaining anxiety. However, this perception could also be (partly) illusory and detached from actual physiology. This dissociation can be assessed in signal detection tasks using the response bias index. To separate interoceptive sensitivity and response bias, a new paradigm applies signal detection theory, allowing for a clear determination of how accurately patients perceive cardiac events. Heart rate variability (HRV) is examined as a marker for cardiac events.

In a previous study, exposure therapy had no impact on the sensitivity of heartbeat perception in both groups. However, the observed null effect could have been caused by neglecting the distinction between interoceptive sensitivity and response bias. In this context, a liberal response strategy has been proposed as a "better safe than sorry" strategy, which can be associated with various psychopathologies. Exposure therapy could contribute to reducing the disconnected physiology in heartbeat perception, thus decreasing the liberal response bias by altering the evaluation of body sensations. In this study, agoraphobic patients with panic disorder and control patients with social anxiety disorder undergo the two heartbeat perception tasks, wherein the sensitivity of heartbeat perception before and after standardized cognitive-behavioral therapy is examined. Additionally, a healthy control group is compared with these two groups regarding the mentioned parameters.

The function of different body systems as a maintaining factor of agoraphobia The endocannabinoid system influences the regulation of various physiological, sensory, motor, emotional, behavioral, and cognitive functions. Patients with panic disorder show increased endocannabinoid concentrations in the blood compared to healthy individuals. How the endocannabinoid system affects the outcome of psychotherapy or is influenced by it remains unclear and will be investigated in the planned study.

The endocannabinoid system modulates the regulation of the Hypothalamic-Pituitary-Adrenal (HPA) axis. Endocannabinoid release acts to inhibit HPA axis activity, reducing cortisol release under acute stress. Reduced cortisol release under acute stress has been observed in PD patients, and this cortisol release has been linked to therapy outcomes. The HPA axis also influences the immune system and cytokine release. Research has shown the impact of anti-inflammatory cytokines (IL-10) on the avoidance behavior of panic patients post-therapy. Thus, the reactivity of the HPA axis and the immune system influence therapy outcomes and predict the success of therapy. Whether therapy influences these body systems and potentially contributes to the normalization of these systems is currently unclear and will be examined in this study. Through the investigation of the HPA axis, as well as the immune and endocannabinoid systems, insights into the interplay of these body systems in panic patients will be gained.

ELIGIBILITY:
Inclusion Criteria:

* Experimental group: Diagnosis of agoraphobia with or without panic disorder
* Clinical control group: diagnosis of social phobia
* Control group: healthy individuals without acute or chronic mental illness
* A depressive disorder may be present as a comorbid diagnosis in the experimental group and the clinical control group

Exclusion Criteria:

* Other mental illnesses: Substance dependence, schizophrenia, bipolar disorder, dementia, eating disorders, PTSD, major depressive episode, personality disorder
* Somatic diseases: Cancer, cardiovascular diseases, epilepsy, autoimmune diseases, metabolic or endocrine diseases
* Taking psychotropic medication (except antidepressants) or medication that affects the cardiovascular system (e.g. beta-blockers), medication containing cortisone, use of creams with corticosteroids
* Pregnancy, breastfeeding
* Ongoing psychotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Extent of Interoceptive Attention | through study completion, an average of 2 years
  Interoceptive attention assessed via a questionnaires (interoceptive attention/ IA). Higher scores reflect a higher interoceptive attention.
Extent of Interoceptive Accuracy | through study completion, an average of 2 years
  Interoceptive accuracy assessed via a questionnaire (interoception accuracy scale/IAS). Higher scores reflect a more accurate/sensitive interoception.
Extent of Objective Interoceptive Sensitivity | through study completion, an average of 2 years
  Interoceptive sensitivity assessed via heart rate measures.
Concentration of Bioparameters under rest and under acute stress | through study completion, an average of 2 years
  Blood measures of cortisol, immune parameters (IL-6, IL-10), endocannabinoids will be assessed under rest and under acute stress during a Trier Social Stress Test. Unit of measure for all biomarkers is pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Petrowski, Prof,, Study Chair — University Medical Center of the Johannes Gutenberg University Mainz
Locations (1):
- University Medical Center, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wittchen HU, Jacobi F, Rehm J, Gustavsson A, Svensson M, Jonsson B, Olesen J, Allgulander C, Alonso J, Faravelli C, Fratiglioni L, Jennum P, Lieb R, Maercker A, van Os J, Preisig M, Salvador-Carulla L, Simon R, Steinhausen HC. The size and burden of mental disorders and other disorders of the brain in Europe 2010. Eur Neuropsychopharmacol. 2011 Sep;21(9):655-79. doi: 10.1016/j.euroneuro.2011.07.018. PMID 21896369
- [Background] Jakubczyk A, Skrzeszewski J, Trucco EM, Suszek H, Zaorska J, Nowakowska M, Michalska A, Wojnar M, Kopera M. Interoceptive accuracy and interoceptive sensibility in individuals with alcohol use disorder-Different phenomena with different clinical correlations? Drug Alcohol Depend. 2019 May 1;198:34-38. doi: 10.1016/j.drugalcdep.2019.01.036. Epub 2019 Mar 8. PMID 30877955
- [Background] Schandry R. Heart beat perception and emotional experience. Psychophysiology. 1981 Jul;18(4):483-8. doi: 10.1111/j.1469-8986.1981.tb02486.x. No abstract available. PMID 7267933
- [Background] Pohl A, Hums AC, Kraft G, Koteles F, Gerlach AL, Witthoft M. Cardiac interoception: A novel signal detection approach and relations to somatic symptom distress. Psychol Assess. 2021 Aug;33(8):705-715. doi: 10.1037/pas0001012. Epub 2021 Apr 8. PMID 33829843
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Griebel G, Stemmelin J, Scatton B. Effects of the cannabinoid CB1 receptor antagonist rimonabant in models of emotional reactivity in rodents. Biol Psychiatry. 2005 Feb 1;57(3):261-7. doi: 10.1016/j.biopsych.2004.10.032. PMID 15691527
- [Background] Kudielka BM, Buske-Kirschbaum A, Hellhammer DH, Kirschbaum C. HPA axis responses to laboratory psychosocial stress in healthy elderly adults, younger adults, and children: impact of age and gender. Psychoneuroendocrinology. 2004 Jan;29(1):83-98. doi: 10.1016/s0306-4530(02)00146-4. PMID 14575731
- [Background] Petrowski K, Herold U, Joraschky P, Wittchen HU, Kirschbaum C. A striking pattern of cortisol non-responsiveness to psychosocial stress in patients with panic disorder with concurrent normal cortisol awakening responses. Psychoneuroendocrinology. 2010 Apr;35(3):414-21. doi: 10.1016/j.psyneuen.2009.08.003. Epub 2009 Nov 12. PMID 19913360
- [Background] Renner V, Conrad R, Kirschbaum C, Lorenz T, Petrowski K. Preliminary results of anti-inflammatory cytokine concentrations predicting therapy outcome in panic disorder. Compr Psychoneuroendocrinol. 2024 Feb 12;17:100227. doi: 10.1016/j.cpnec.2024.100227. eCollection 2024 Feb. PMID 38404508
- [Background] Wechsler TF, Kumpers F, Muhlberger A. Inferiority or Even Superiority of Virtual Reality Exposure Therapy in Phobias?-A Systematic Review and Quantitative Meta-Analysis on Randomized Controlled Trials Specifically Comparing the Efficacy of Virtual Reality Exposure to Gold Standard in vivo Exposure in Agoraphobia, Specific Phobia, and Social Phobia. Front Psychol. 2019 Sep 10;10:1758. doi: 10.3389/fpsyg.2019.01758. eCollection 2019. PMID 31551840